CLINICAL TRIAL: NCT01673685
Title: Randomised Crossover Trial of Portable Oxygen Cylinders Versus Battery Powered Portable Oxygen Concentrators
Brief Title: Trial of Portable Oxygen Cylinders Versus Battery Powered Portable Oxygen Concentrators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Kristin Carson, Research Scientist, The Queen Elizabeth Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010090
Record Dates: First submitted 2012-08-15; First posted 2012-08-28 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: COPD
Keywords: COPD; Oxygen cylinder; Portable oxygen cylinder; Battery powered delivery device; mobility; dyspnoea; Quality of Life; Cost effectiveness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: Portable oxygen concentrators vs oxygen cylinders
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Portable Oxygen Cylinder (Placebo Comparator): Portable Oxygen Cylinder
  Interventions: Device: Portable Oxygen
- Portable Oxygen Concentrator (Active Comparator): Portable Oxygen Concentrator
  Interventions: Device: Portable Oxygen

INTERVENTIONS:
Device: Portable Oxygen
  Other Names: Respironics Airsep (rental) AssetNumber 38269

SUMMARY:
Randomised cross-over study of portable oxygen concentrators compared to oxygen cylinders to improve quality of life and other outcomes for patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Many patients with Chronic Obstructive Pulmonary Disease (COPD) have limited activities of daily living (shopping, visiting friends, going for a walk) due to exertional dyspnoea. State Government funding provides up to 4 oxygen cylinders to be delivered to patients requiring portable oxygen per month. However, the more active and motivated COPD patients often find these gratis supplies run out well before the month is up. Recent technology has developed battery powered portable oxygen concentrators. The latest models weigh less than a typical oxygen cylinder and have the advantage that the battery plug can be plugged into a car cigarette lighter outlet, or into the power point of any house. This means that the COPD patient has the potential to be far more mobile for far longer periods of time and visit friends almost infinitely by recharging the battery pack during the course of their travels. The latest battery powered oxygen device weighs 2kgs which is about half that of an oxygen cylinder. However, there is an upfront expense to these devices and inevitably a sound business case with cost considerations (amortization of the initial purchase price, recharging the battery costing the patient's electricity etc) needs consideration. Also, before assuming these devices are superior (or at least as good as) oxygen cylinders, because they have a pulsed delivery of oxygen technology i.e. the oxygen is delivered in bursts with each inspiration that is detected, unlike oxygen cylinders which can run continuously, one cannot assume without rigorous evaluation that mobility and quality of life necessarily is good or superior with the new devices. Hence, quality of life evaluation with emphasis on enjoyed activities by each COPD patient are essential as well as costing issues for the funding stakeholder (i.e. hospital site specific funds). Should a sound business case be made (i.e. improved quality of life with less costs over a longer period of time), then a sound justification can be made to funding bodies that COPD patients are better off and the funding body is shouldering less cost by wider usage of these devices following evaluation of this project. The design will be a randomised crossover such that COPD patients will spend one month on oxygen or battery powered concentrator devices and then switch over to the other oxygen delivery. Chronic Respiratory Questionnaire (Quality of Life) will be administered at the end of each month.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients diagnosed with stable COPD
* currently prescribed and using portable oxygen cylinders with a "pulsed" oxygen delivery for exertion.

Exclusion Criteria:

* Co-morbidities such as: other major respiratory conditions, cardiac or other substantial co-morbidities which significantly limit mobility independent of COPD
* Baseline step test which demonstrates a reduced effect on the battery device compared to oxygen cylinders.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Quality of life as measured through Chronic Respiratory Questionnaire | One month
  only two subdomains of the Chronic Respiratory Questionnaire (CRQ) were used: the Shortness of Breath (SoB) domain and the Mastery domain

SECONDARY OUTCOMES:
Patient Preference | One month
  Five 7-point Likert Scales, ranging from 1 (none of the time) to 7 (all of the time) on portability ("the equipment was portable enough for my needs"), operation ("I was able to set up and operate the equipment properly"), noise ("Noise from the equipment affected me"), comprehension ("I was able to understand the functions of the equipment, e.g. alarms") and duration ("The oxygen lasted long enough for me to perform my normal activities"). Furthermore, patients were asked to provide comments on use of the POCs and the Cylinders after they completed the respective stage of the trial.
Cost effectiveness of portable oxygen concentrator compared to cylinder | one month
  Economic assessment based on treatment cost, readmission data and hospital utilisation
Quality of life as measured through AQoL-8D | One month
  Assessment of Quality of Life (AQoL)-8D Multi-Attribute Utility Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Smith, MBBS, FRACP, PhD, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- The Queen Elizabeth Hospital, Woodville Road, Woodville, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon request.